CLINICAL TRIAL: NCT03451565
Title: Intraoperative Systemic Arterial Hypotension Secondary to Beach Positioning : an Observational Study
Brief Title: Intraoperative Systemic Arterial Hypotension Secondary to Beach Positioning
Acronym: HypoTAShoulder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7009
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-02

CONDITIONS: Hypotension
Keywords: Hypotension; Systemic blood pressure
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at describing the systemic arterial hypotension secondary to intraoperative beach chair positioning. This is a non-interventional prospective study.

The primary endpoint will be the intraoperative systemic arterial pressure measured at the arm.

The secondary endpoints will include postoperative mortality, intensive care admission, post anesthesia care unit length of stay,

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Patient operated in a sitting position at Hopitaux Universitaires de Strasbourg
* Patient willing to participate in the study

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied will include patients operated at the University Hospitals of Strasbourg in a sitting position.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 10 min after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eric Noll, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service D'Anesthesiologie - Reanimation Chirurgicale, Strasbourg, France